CLINICAL TRIAL: NCT06697613
Title: Development and Validation of a Prediction Model for Acute Kidney Injury Following Cisplatin-Based HIPEC in Patients With Ovarian Cancer: a Multi-center Retrospective Cohort Study
Brief Title: Development and Validation of a Prediction Model for AKI Following Cisplatin-Based HIPEC in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Jing Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-959-01
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; AKI - Acute Kidney Injury
MeSH Terms: conditions — Ovarian Neoplasms; Acute Kidney Injury | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRS-HIPEC
  Interventions: Procedure: Hyperthermic intraperitoneal chemotherapy

INTERVENTIONS:
Procedure: Hyperthermic intraperitoneal chemotherapy — Patients diagnosed with FIGO Stage 3 or stage 4 ovarian cancer received hyperthermic intraperitoneal chemotherapy with cisplatin following cytoreductive surgery including primary debulking surgery, interval debulking surgery and secondary debulking surgery.

SUMMARY:
Ovarian cancer is the most lethal malignant tumor of the female reproductive system. Cytoreduction surgery(CRS) combined with chemotherapy is the primary method for treating ovarian cancer, and complete tumor resection is an important means to improve prognosis. It has been demonstrated that the use of cisplatin for hyperthermic intraperitoneal chemotherapy (HIPEC) following CRS can significantly improve the prognosis of some patients with ovarian cancer. However, HIPEC with cisplatin can lead to acute kidney injury (AKI), a serious complication that can seriously affect the patient's short- and long-term prognosis. NCCN guidelines recommend the use of sodium thiosulfate in all patients receiving HIPEC. This study intends to retrospectively collect clinical characteristics of patients to establish a prediction model for kidney injury, with a view to screening those at high risk of kidney injury for use of sodium thiosulfate for nephrotoxicity rescue in cisplatin HIPEC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received HIPEC with cisplatin following cytoreductive surgery.
* Patients diagnosed with ovarian cancer pathologically.
* FIGO stage III-IV.

Exclusion Criteria:

* Use of renal protective drugs such as sodium perthiosulfate.
* Any grade of chronic or acute renal disease or other serious complications existed before HIPEC.
* Patients with single kidney.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ovarian cancer were treated with cytoreductive surgery combined with hyperthermic intraperitoneal chemotherapy with cisplatin.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Model prediction Probability | Up to 7 days within CRS-HIPEC
  Using the constructed clinical prediction model, the patient's baseline characteristics were input, and the model would output the probability of the patient developing AKI.
AUC (Area Under Curve) | Up to 7 days within CRS-HIPEC
  The AUC value of the model was calculated using the ROC (Receiver Operating Characteristic) Curve.

SECONDARY OUTCOMES:
The incidence of AKI. | Up to 7 days within CRS-HIPEC
  The AKI would be diagnosed according to KDIGO 2012 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Colombo N, Sessa C, du Bois A, Ledermann J, McCluggage WG, McNeish I, Morice P, Pignata S, Ray-Coquard I, Vergote I, Baert T, Belaroussi I, Dashora A, Olbrecht S, Planchamp F, Querleu D; ESMO-ESGO Ovarian Cancer Consensus Conference Working Group. ESMO-ESGO consensus conference recommendations on ovarian cancer: pathology and molecular biology, early and advanced stages, borderline tumours and recurrent diseasedagger. Ann Oncol. 2019 May 1;30(5):672-705. doi: 10.1093/annonc/mdz062. PMID 31046081
- [Background] Zivanovic O, Chi DS, Filippova O, Randall LM, Bristow RE, O'Cearbhaill RE. It's time to warm up to hyperthermic intraperitoneal chemotherapy for patients with ovarian cancer. Gynecol Oncol. 2018 Dec;151(3):555-561. doi: 10.1016/j.ygyno.2018.09.007. Epub 2018 Sep 22. PMID 30249527
- [Background] Lemoine L, Sugarbaker P, Van der Speeten K. Drugs, doses, and durations of intraperitoneal chemotherapy: standardising HIPEC and EPIC for colorectal, appendiceal, gastric, ovarian peritoneal surface malignancies and peritoneal mesothelioma. Int J Hyperthermia. 2017 Aug;33(5):582-592. doi: 10.1080/02656736.2017.1291999. PMID 28540826
- [Background] Hod T, Freedberg KJ, Motwani SS, Chen M, Frendl G, Leaf DE, Gupta S, Mothi SS, Richards WG, Bueno R, Waikar SS. Acute kidney injury after cytoreductive surgery and hyperthermic intraoperative cisplatin chemotherapy for malignant pleural mesothelioma. J Thorac Cardiovasc Surg. 2021 Apr;161(4):1510-1518. doi: 10.1016/j.jtcvs.2020.05.033. Epub 2020 May 29. PMID 32631662